CLINICAL TRIAL: NCT05531578
Title: Transfemoral Implant of Inovare® Transcatheter Valve - Clinical Trial of Feasibility and Safety and Efficacy Verification
Brief Title: Transfemoral Implant of Inovare® Transcatheter Valve
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Braile Biomedica Ind. Com. e Repr. Ltda. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Inovare - Transfemoral
Record Dates: First submitted 2022-08-18; First posted 2022-09-08 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Aortic Valve Stenosis
Keywords: TAVI; TAVR; Transfemoral; Transcatheter Valve
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TAVI TRANSFEMORAL (Experimental)
  Interventions: Device: INOVARE® Transcatheter Valve, NexusCath Delivery System, Aureus Expandable Introducer, Balloon Catheter for Pre-Dilation and Compression Device (Crimper)

INTERVENTIONS:
Device: INOVARE® Transcatheter Valve, NexusCath Delivery System, Aureus Expandable Introducer, Balloon Catheter for Pre-Dilation and Compression Device (Crimper) — Transfemoral implantation of the INOVARE® transcatheter valve

SUMMARY:
Clinical trial to evaluate the early safety and efficacy of the transfemoral implant of Inovare® Transcatheter Valve for the treatment of patients with severe degenerative aortic stenosis and high surgical risk.

DETAILED DESCRIPTION:
The Inovare® transcatheter valve was developed and has been market ed since 2011 for replacement, via transapical or transaortic route, of calcified native aortic valves and degenerated bioprostheses (aortic and mitral) with satisfactory medium-long-term results. The present study aims to evaluate the safety and clinical performance of the new navigation and delivery system of this device using the transfemoral route. The new device has as its main feature the drivable control of the curvature of the delivery system, the which allows better navigability in regions of more complex anatomy, especially with accentuated tortuosities.

ELIGIBILITY:
Inclusion Criteria:

* Calcified degenerative aortic stenosis with valve area < 1.0 cm2 (or valve area index < 0.6 cm2/m2) and mean transvalvular gradient > 40 mmHg or aortic jet velocity > 4 m/s by echocardiogram.
* Multidisciplinary evaluation by the "Heart Team", composed of a cardiovascular surgeon, clinical cardiologist and hemodynamicist, which concludes that the patient has:

  * High surgical risk for aortic valve replacement, typically with an STS score of ≥ 8% (or logistic EuroSCORE ≥ 20%) or intermediate risk (STS of ≥ 3% and < 8%);
  * Presence of porcelain aorta or hostile chest, as well as global clinical condition and comorbidities not fully addressed by the score STS
  * Presence of extreme frailty (5-meter walk test [5MWT], grip strength, activities of daily living (ADL), and albumin laboratory exam);
  * Considerable chance of clinical benefit with the transcatheter procedure.
* Heart failure symptoms NYHA functional ≥ II.
* Aortic valve annulus with a mean diameter between 17.3 and 28.6 mm, documented by imaging method, suitable for positioning and accommodation of the Inovare® prosthesis, according to the judgment of an experienced hemodynamicist.
* Height of coronary ostia > 10 mm or presence of a coronary graft that prevents the occurrence of acute myocardial ischemia due to coronary occlusion after valve release.
* Femoral arterial access route considered adequate for the progression of the vascular introducer and prosthesis-balloon system, typically evaluated through multi-imaging methods that include, for example, conventional angiography and computed tomography.
* Patient has provided written informed consent to participate in the trial.

Exclusion Criteria:

Clinic

* Hemodynamic instability requiring vasoactive drugs or circulatory support;
* Valve procedure with clinical need to be performed in a time of urgency or emergency (non-elective);
* Left ventricular ejection fraction < 30%;
* Chronic renal failure on dialysis or with serum creatinine levels > 3.0 mg/dL (265 µmol/L);
* Acute renal failure with serum creatinine that has not yet returned to baseline levels;
* Clinical or biological signs of infection with systemic repercussions;
* Endocarditis < 12 months;
* Coronary artery disease requiring elective revascularization during or after the valve procedure;
* Evidence of myocardial infarction in an interval of less than one month;
* Recent stroke or transient ischemic attack (within the last 6 months);
* Hypersensitivity or contraindication to the administration of heparin, ticlopidine or clopidogrel or to radiopaque contrast;
* Anemia (hemoglobin < 10 g/dl), thrombocytopenia (< 100,000 cells/mm3) or hyperthrombocytosis (> 700,000 cells/mm3);
* Need for chronic anticoagulation for other causes;
* Active peptic disease, gastrointestinal bleeding < 3 months, or previously diagnosed bleeding diathesis;
* Life expectancy less than 12 months due to non-cardiac disease or other comorbidities.

Anatomical/morphological

* Valve ring diameter less than or equal to 17.2 mm or greater than or equal to 28.7 mm;
* Iliofemoral access route, with extreme tortuosity or calcification or reduced luminal diameter (typically < 7 mm), which prevents safe progression of the arterial introducer and delivery system with the prosthesis, according to the judgment of the responsible physician;
* Presence of sessile and unstable atheromas in the ascending aorta and/or aortic arch detected by imaging methods;
* Obstructive hypertrophic cardiomyopathy or severe left ventricular outflow tract obstruction, with no possibility of balloon dilation;
* Previous aortic or mitral valve procedure (surgical or by catheter, excluding aortic balloon valvuloplasty);
* Moderate or severe aortic, mitral or tricuspid regurgitation;
* Non-calcified native valve;
* Evidence of an intracardiac mass (tumor, thrombus, or vegetation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-09-11 (Actual); Primary Completion 2024-02-20 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Device success | Procedure
  Absence of mortality in the procedure AND correct positioning of a single bioprosthesis with the intended performance (mean gradient < 20 mmHg and regurgitation ≥ moderate).
Death the first 30 days | 30 days
  Deaths from any cause within the first 30 days of the procedure or during hospital stay will be considered procedure-related deaths.

SECONDARY OUTCOMES:
Device success | 30 days or more
  Absence of mortality in the procedure AND correct positioning of a single bioprosthesis with the intended performance (mean gradient < 20 mmHg and regurgitation ≥ moderate).
Incidence of serious adverse events | 30 days or more
  Overall mortality; · Coronary obstruction requiring percutaneous intervention (PCI); · Stroke; · Stage 2-3 acute kidney injury requiring dialysis technique or increase in creatinine ≥ 300% or creatinine ≥4.0 mg/dl; · Life-threatening bleeding (or sequelae) or critical organ bleeding or hypovolemic shock or severe hypotension requiring vasopressors or surgery or packed red blood cells (RBCs) transfusion ≥4 units; · Major vascular complication; · Reintervention for valvular dysfunction; · Myocardial infarction; ·Permanent pacemaker implantation
Efficacy of the procedure | 30 days or more
  Mortality, stroke, bioprosthesis dysfunction due to stenosis (mean gradient ≥ 20 mmHg) and regurgitation ≥ moderate, re-hospitalization with congestive heart failure or valvular symptoms, New York Heart Association (NYHA) functional class III or IV.

CONTACTS AND LOCATIONS:
Overall Officials: José Honório de Almeida Palma da Fonseca, Dr, Principal Investigator — InCor Heart Institute
Locations (4):
- Brazil (4):
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, São José do Rio Preto
  - INCOR - Instituto do Coração do Hospital das Clínicas da FMUSP, São Paulo
  - Instituto Dante Pazzanese de Cardiologia, São Paulo
  - Universidade Federal de São Paulo, São Paulo